CLINICAL TRIAL: NCT00494494
Title: Effect of Nepafenac on Post-operative Cystoid Macular Edema Following Uncomplicated Cataract Surgery
Brief Title: Effect of Nepafenac on Post-operative Macular Swelling Following Uncomplicated Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Research to Prevent Blindness (Other)
Responsible Party: Kenneth Cohen, MD, UNC Chapel Hill
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-3115
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Cystoid Macular Edema
Keywords: cystoid macular edema; cataract; nonsteroidal antiinflammatory drugs; optical coherence tomography
MeSH Terms: conditions — Macular Edema; Cataract | interventions — Standard of Care; nepafenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (Active Comparator): topical antibiotic for 10 days and a topical corticosteroid for 1 month
  Interventions: Drug: Standard Care
- Nepafenac (Experimental): 1 drop per study eye three times per day for 30 days in addition to standard care
  Interventions: Drug: nepafenac

INTERVENTIONS:
Drug: Standard Care — topical antibiotic for 10 days plus topical corticosteroids for 1 month
  Arms: Standard Treatment
Drug: nepafenac — liquid drops, administered three times per day for 1 month in addition to standard care use of topical antibiotic and topical corticosteroid
  Arms: Nepafenac

SUMMARY:
Purpose: Study the effect of nepafenac ophthalmic suspension 0.1% to prevent post-operative cystoid macular edema following uncomplicated cataract surgery

Participants: Patients having cataract surgery at UNC who meet eligibility criteria

Procedures (methods): Patients will have pre and post-operative vision measured and optical coherence tomography (OCT) testing, also cataract density and intraoperative phacoemulsification parameters including ultrasound power and ultrasound time will be measured. Patients will be randomized into two groups. Group 1 will be treated with standard post-operative cataract management. Group 2 will be treated with standard post-operative cataract management plus topical nepafenac for one month. Post-operative macular thickness will be studied by analyzing the visual acuity and OCT measurements at two months post surgery.

DETAILED DESCRIPTION:
We plan to enroll 80 patients in this prospective randomized clinical trial. Eligible patients will be randomized into two groups. All patients will have pre-operative Early Treatment of Diabetic Retinopathy Study (ETDRS) vision measured and pre-operative OCT (Humphrey-Zeiss Medical Systems, San Leandro, CA) in both eyes. OCT measurements will include total macular volume, central foveal thickness, and average macular thickness. Pre-operatively, all cataracts will be graded using the LOCS III classification system.10 Group 1 will receive pre-operative topical nepafenac to maintain intra-operative pupillary dilation which is standard care for cataract surgery. Following surgery Group 1 will be treated with standard post operative cataract treatment, including a topical antibiotic and a topical corticosteroid. Group 2 will also receive pre-operative topical nepafenac to maintain intra-operative pupillary dilation. Following surgery patients in Group 2 will be treated with topical nepafenac, a topical antibiotic, and a topical corticosteroid. Group 2 will be given the 3ml bottle of nepafenac to take home and instructed to use it three times per day for one month. Intra-operative surgical parameters including ultrasound time and average percent phacoemulsification power will be recorded for all surgeries. All patients will be seen on post-operative day one, one week, one month, and two months. At the two month visit, best corrected ETDRS vision and OCT will be repeated in both eyes. The two month visual acuity and post-operative OCT will be analyzed to evaluate the effect of nepafenac on CME following cataract surgery. Wilcoxon signed rank test will be used to compare pre-operative and post-operative differences between visual acuity and OCT measurements. The Spearman correlation will be used to compare the variables in the study including cataract density, ultrasound time, average percent phacoemulsification power, and OCT measurements.

ELIGIBILITY:
Inclusion Criteria:

* over age 50
* having cataract surgery at UNC

Exclusion Criteria:

* medically controlled diabetes
* history of intraocular surgery
* abnormal pre-op optical coherence tomography scan
* history of ocular inflammation
* have age related macular degeneration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Cohen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: These subjects only received the standard of care for post-operative cataract, which consists of a topical antibiotic and a topical corticosteroid.
- Nepafenac: 1 drop per study eye three times per day for 30 days plus standard care
Period: Overall Study
Arm/Group | Standard Treatment | Nepafenac
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Nepafenac | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 40 | 39 | 79
Age Continuous [Mean (Standard Deviation); unit: years] | 70.33 (8.04) | 73.95 (8.99) | 72.14 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Central Macular Thickness (Difference in Mean Pre-post Changes by the Two Treatment Groups)
Description: The endpoints of the study were change in macular thickness measured by OCT in the central 1mm diameter centred on the fovea (central macular thickness)
Time Frame: baseline and 8 weeks
Population: Three subjects in the treatment group and two subjects in the control group had unreliable preoperative OCT scans because of dense posterior subcapsular cataracts. These subjects were excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Standard Treatment | Nepafenac
Number analyzed (Participants) | 40 | 39
microns | 2.78 [-10.12 to 15.68] | 5.6 [-8.2 to 19.4]
Statistical Analysis 1: Comparison: Standard Treatment vs Nepafenac; The null hypothesis is that there is no correlation between the 2 groups. Standard methods were used for power calculation to determine the sample size needed to have 0.90 power for the comparison between two groups at the two-sided significance of 0.05; Test type: Non-Inferiority or Equivalence — Our estimate of a clinically relevant increase is 25 microns. With these specifications, the sample size that is required to have 0.90 power for the comparison between two groups at the two-sided 0.05 significance level is about 10 per group; p = 0.7029, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.82, 95% CI 2-sided [-3.27 to 8.91], Standard Deviation 13.8

2. Primary Outcome: Pre-operative Best Corrected Visual Acuity (BCVA)
Description: Patients were instructed to read letters on the EDTRS visual acuity chart. The mean and standard deviation for each group was measured. Letters range from 0 (20/2000) to 110 (20/12.5), with the higher number signaling better visual acuity.
Time Frame: baseline
Population: The analysis was per protocol. At baseline, everybody was given a Best Corrected Visual Acuity Assessment (BCVA).
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Standard Treatment | Nepafenac
Number analyzed (Participants) | 40 | 39
letters | 38.48 (9.83) | 40.49 (9.56)
Statistical Analysis 1: Comparison: Standard Treatment vs Nepafenac; Test type: Superiority or Other; p = 0.1937, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.01, 95% CI 2-sided [-2.41 to 6.43], Standard Deviation 9.56

3. Primary Outcome: Foveal Thickness
Description: difference in mean pre-post changes by the two treatment groups
Time Frame: baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Standard Treatment | Nepafenac
Number analyzed (Participants) | 40 | 39
microns | -2.0 [-25.4 to 21.4] | 4.7 [-14.9 to 24.3]
Statistical Analysis 1: Comparison: Standard Treatment vs Nepafenac; Test type: Superiority or Other; p = 0.5066, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 6.70, 95% CI 2-sided [-3.12 to 16.52], Standard Deviation 19.6

4. Primary Outcome: Macular Volume (Difference in Mean Pre-post Changes by the Two Treatment Groups)
Time Frame: baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Standard Treatment | Nepafenac
Number analyzed (Participants) | 40 | 39
microns | 0.05 [-0.46 to 0.56] | 0.10 [-0.11 to 0.31]
Statistical Analysis 1: Comparison: Standard Treatment vs Nepafenac; Test type: Superiority or Other; p = 0.5099, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.13 to 0.227], Standard Deviation 0.21

5. Primary Outcome: Post-operative Best Corrected Visual Acuity (BCVA)
Description: The patients were again instructed to read letters on the ETDRS chart 8 weeks post-surgery. The mean and standard deviation for each group was recorded. Letters range from 0 (20/2000) to 110 (20/12.5), with the higher number signaling better visual acuity.
Time Frame: baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: letters
Arm/Group | Standard Treatment | Nepafenac
Number analyzed (Participants) | 40 | 39
letters | 54.46 [39 to 67] | 55.49 [44 to 65]
Statistical Analysis 1: Comparison: Standard Treatment vs Nepafenac; Test type: Superiority or Other; p = 0.5005, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.03, 95% CI 2-sided [-1.49 to 3.55], Standard Deviation 5.64

ADVERSE EVENTS:
Description: Serious and/or other adverse Events were not collected for this study.
Arm/Group | Standard Treatment | Nepafenac
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Although the peak incidence of CME is said to be at 4-12 weeks after surgery, we may have missed the time course for detecting the maximum increased OCT measured macular thickness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes